CLINICAL TRIAL: NCT03013556
Title: A Prospective, Randomized, Multicenter, Open-label Study of Optimal Antiviral Treatment in HBeAg Positive Chronic Hepatitis B Patients
Brief Title: Study on an Optimal Antiviral Treatment in HBeAg Positive Chronic Hepatitis B Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Xinxin Zhang, vice president of Ruijin hospital(North collegue), Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHDC12016101
Record Dates: First submitted 2016-12-16; First posted 2017-01-06 (Estimated); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Chronic Hepatitis
Keywords: HBeAg positive
MeSH Terms: conditions — Hepatitis, Chronic | interventions — Tenofovir; peginterferon alfa-2a

ARMS (3):
- Group A,TDF (Active Comparator): The subjects in group A will be treated by TDF for 96 weeks
  Interventions: Drug: Group A, TDF
- Group B,TDF+PEG (Experimental): The subjects in group B will be treated by TDF in the first 48 weeks, then will be treated by the combination of TDF and Peginterferon alfa-2a for another 48 weeks
  Interventions: Drug: Group B:TDF then TDF and Peginterferon alfa-2a
- Group C,TDF+PEG (Experimental): The subjects in group C will be treated by the combination of TDF and Peginterferon alfa-2a for the first 48 weeks, then will be treated by TDF for another 48 weeks
  Interventions: Drug: Group C:TDF and Peginterferon alfa-2a then TDF

INTERVENTIONS:
Drug: Group A, TDF — TDF for 96 weeks
  Other Names: tenofovir
  Arms: Group A,TDF
Drug: Group B:TDF then TDF and Peginterferon alfa-2a — Subjects will be treated by TDF in the first 48 weeks, then will be treated by the combination of TDF and Peginterferon alfa-2a for another 48 weeks
  Other Names: tenofovir,pegasys
  Arms: Group B,TDF+PEG
Drug: Group C:TDF and Peginterferon alfa-2a then TDF — Subjects will be treated by the combination of TDF and Peginterferon alfa-2a for the first 48 weeks, then will be treated by TDF for another 48 weeks.
  Other Names: tenofovir,pegasys
  Arms: Group C,TDF+PEG

SUMMARY:
The current study is a prospective, randomized, open, multi-center investigation. The aim of the study is to investigate whether the HBeAg seroconversion rate can be improved if applying combination therapy in HBeAg positive CHB patients who has achieved HBVDNA<105copies/ml，HBsAg≤5000IU/ml, ALT≥ 2ULN or Liver histology G2S2.

DETAILED DESCRIPTION:
The HBeAg positive chronic hepatitis B(CHB) subjects who has achieved HBV DNA<10*5copies/ml，HBsAg≤5000IU/ml, ALT≥ 2ULN or Liver histology G2S2 will be randomized to three groups. The subjects who go into group A will be treated by tenofovir disoproxil fumarate (TDF) for 96 weeks; The subjects who go into group B will be treated by TDF in the first 48 weeks, then will be treated by the combination of TDF and Peginterferon alfa-2a for another 48 weeks; The subjects who go into group C will be treated by the combination of TDF and Peginterferon alfa-2a for the first 48 weeks, then will be treated by TDF for another 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients with age ≥18 and ≤65 years;
2. There should be evidences that HBsAg and HBeAg have been positive for more than 6 months with HBsAb and HBeAb negative;HBsAg≤50000IU/ml, ALT≥ 2ULN,Liver histology above G2S2 and HBV DNA≥10*5 copies/mL;
3. Women without ongoing pregnancy or breast feeding and both women and men willing to take an effective contraceptive measure during the treatment;
4. Agree to participate in the study and sign the patient informed consent form.

Exclusion Criteria:

1. Treated by immunosuppressant,immunomodulator,Systemic cytotoxic drug,herbs or HBIg within 6 months prior to the first dose of treatment;
2. ALT≥10 X ULN or total bilirubin ≥2 X ULN;
3. Allergic history to interferon;
4. Co-infection with active hepatitis A, hepatitis C, hepatitis D and/or human immunodeficiency virus (HIV);
5. Child-Pugh scores >7;
6. History or other evidence of a medical condition associated with chronic liver disease other than viral hepatitis (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures, thalassemia);
7. Pregnant or breast-feeding Women;
8. Consuming alcohol in excess of 20g/day for women and 30g/day for men within 6 months prior to enrollment or drug taking history;
9. ANC(absolute neutrophil count)<1.5x 10^9/L or PLT(platelet count)<90x 10^9/L
10. Creatinine over upper limit of normal;
11. History of severe psychiatric disease, especially depression. Severe psychiatric disease is defined as major depression or psychosis that treated with antidepressant medication or a major tranquilizer at therapeutic doses respectively at any time prior to 3 months or any history of the following: a suicidal attempt hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease;
12. History of immunologically mediated disease, (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, scleroderma, rheumatoid arthritis etc.);
13. History of esophageal varices bleeding or other evidence of esophageal varices bleeding or other symptoms consistent with decompensated liver disease;
14. History of severe cardiac disease (e.g., New York Heart Association Functional Class III or IV, myocardial infarction within 6 months, ventricular tachyarrhythmias requiring ongoing treatment, unstable angina or other significant cardiovascular diseases);
15. Hemodialysis patients or patients with renal insufficiency;
16. History of a severe seizure disorder or current anticonvulsant use;
17. Major organ transplantation or other evidence of severe illness, malignancy, or any other conditions, which would make the patient, in the opinion of the investigator, unsuitable for the study;
18. History of thyroid disease poorly controlled on prescribed medications;
19. Evidence of severe retinopathy or clinically relevant ophthalmologic disorder;
20. History of other severe disease or evidence of other severe disease or any other illness or conditions that the investigator believe that patients are not suitable to join in the study;
21. Patients included in another trial or having been given investigational drugs within 12 weeks prior to screening;
22. AFP(alpha feto protein)>50ng/ml and/or evidence of hepatocellular carcinoma;
23. Other disease should exclusive considered by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2016-11; Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of subjects who achieve HBeAg seroconversion | at 96 week
  The number of subjects with HBeAg seroconversion at week 96 will be measured

SECONDARY OUTCOMES:
Number of participants who achieve HBeAg seroconversion | at 48 week;at 72 week
  The number of subjects with HBeAg seroconversion at week 48 and 72 will be measured
The percentage decrease of HBsAg level at group A,B,C | at 48 week;at 72 week;at 96 week
  The level of HBsAg in group A,B,C at week 48 ,72 and 96 will be measured,changing from baseline
Number of participants who achieve HBeAg loss | at 48 week;at 72 week;at 96 week
  The number of subjects with HBeAg loss at week48.72 and 96 will be measured
The number of subjects who achieve HBVDNA undetectable | at 24 week;48 week;at 72 week;at 96 week
  The number of subjects with HBVDNA undetectable at week 24,48,72 and 96 will be measured
The factor such as HBsAg level related to responsible rate | at week 48,72,96
  The HBsAg level at week 48,72,96 will be measured, to assess whether the quantitative HBsAg level related to the responsible rate
The number of subjects who achieve ALT back to normal | at 48 week;at 72 week;at 96 week
  The number of subjects with normal ALT at week 48,72 and 96 will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Xinxin Zhang, Principal Investigator — Ruijin Hospital
Locations (8):
- China (8):
  - Xixi Hospital of Hangzhou, Hangzhou
  - Changhai Hospital, Shanghai
  - Hua shan Hospital,Fudan University, Shanghai
  - Infectious diesease hospital of Huangpu district in Shanghai, Shanghai
  - No.9 hospital of shanghai, Shanghai
  - Shanghai public health clinical center, Shanghai
  - Shuguang Hospital of Shanghai T.C.M, Shanghai
  - Tongren hospital Shanghai Jiaotong University School of medicine, Shanghai

REFERENCES:
- [Result] Marcellin P, Ahn SH, Ma X, Caruntu FA, Tak WY, Elkashab M, Chuang WL, Lim SG, Tabak F, Mehta R, Petersen J, Foster GR, Lou L, Martins EB, Dinh P, Lin L, Corsa A, Charuworn P, Subramanian GM, Reiser H, Reesink HW, Fung S, Strasser SI, Trinh H, Buti M, Gaeta GB, Hui AJ, Papatheodoridis G, Flisiak R, Chan HL; Study 149 Investigators. Combination of Tenofovir Disoproxil Fumarate and Peginterferon alpha-2a Increases Loss of Hepatitis B Surface Antigen in Patients With Chronic Hepatitis B. Gastroenterology. 2016 Jan;150(1):134-144.e10. doi: 10.1053/j.gastro.2015.09.043. Epub 2015 Oct 8. PMID 26453773
- [Result] Xie Q, Zhou H, Bai X, Wu S, Chen JJ, Sheng J, Xie Y, Chen C, Chan HL, Zhao M. A randomized, open-label clinical study of combined pegylated interferon Alfa-2a (40KD) and entecavir treatment for hepatitis B "e" antigen-positive chronic hepatitis B. Clin Infect Dis. 2014 Dec 15;59(12):1714-23. doi: 10.1093/cid/ciu702. Epub 2014 Sep 4. PMID 25190434
- [Result] Brouwer WP, Xie Q, Sonneveld MJ, Zhang N, Zhang Q, Tabak F, Streinu-Cercel A, Wang JY, Idilman R, Reesink HW, Diculescu M, Simon K, Voiculescu M, Akdogan M, Mazur W, Reijnders JG, Verhey E, Hansen BE, Janssen HL; ARES Study Group. Adding pegylated interferon to entecavir for hepatitis B e antigen-positive chronic hepatitis B: A multicenter randomized trial (ARES study). Hepatology. 2015 May;61(5):1512-22. doi: 10.1002/hep.27586. Epub 2015 Feb 27. PMID 25348661